CLINICAL TRIAL: NCT02202629
Title: The Effects of Different Combinations of Plant Based Extracts on Cognitive Function and Cerebral Blood Flow in Humans
Brief Title: Plant Based Extracts and Cognition
Acronym: CEOPTB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1406
Record Dates: First submitted 2014-07-24; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Change in Cognitive Function and Fatigue During Extended Performance of the Cognitive Demand Battery (CDB) at 1, 3 and 6 Hours Post Consumption; Change in Long Term Declarative Memory at 1, 3 and 6 Hours Post-intervention.

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cherry flavoured beverage 1 (Placebo Comparator): 10floz cherry flavoured test article
- Cherry flavoured beverage 2 (Experimental): 10floz of cherry flavoured test article with fruit, vegetable and herbal extracts
  Interventions: Other: Beverage containing plant based extracts
- Cherry flavoured beverage 3 (Experimental): 10floz of cherry flavoured test article with fruit, vegetable and herbal extracts
  Interventions: Other: Beverage containing plant based extracts
- Cherry flavoured beverage 4 (Experimental): 10floz of cherry flavoured test article with fruit, vegetable and herbal extracts
  Interventions: Other: Beverage containing plant based extracts

INTERVENTIONS:
Other: Beverage containing plant based extracts — Intervention involves single exposure, oral consumption of test article following baseline measurements
  Arms: Cherry flavoured beverage 2; Cherry flavoured beverage 3; Cherry flavoured beverage 4

SUMMARY:
Acute, randomized, placebo controlled, double blind, 4 arm crossover study to determine the effect of different combinations of plant based extracts on cognitive function and cerebral blood flow.

DETAILED DESCRIPTION:
The objectives of this study are to assess the effects of oral consumption of three differing combinations of plant based extracts, on cognitive function and cerebral blood flow (using Near infrared Spectroscopy) in comparison to placebo. The primary outcome will be change in cognitive function and mental fatigue during extended performance of the Cognitive Demand Battery (CDB) at 1, 3 and 6 hours post- consumption.

ELIGIBILITY:
Inclusion Criteria:

* Are over 18 or under 49 years of age
* Self-report of good health
* Are not excluded on the basis of the following exclusion criteria
* English is first language (some of the cognitive tests have only been validated in native English speakers)

Exclusion Criteria:

* Are below 18 or above 49 years of age
* Are a smoker
* Have food allergies or sensitivities to any of the ingredients contained in the investigational product or any other foodstuff
* Currently take medication except the contraceptive pill
* Have habitually used dietary supplements within the last month (defined as more than 3 consecutive days or 4 days in total)
* Have sleep disturbances and/or are taking sleep aid medication
* Have a Body Mass Index (BMI) outside of the range 18-35 kg/m2
* Have high blood pressure (systolic over 139 mm Hg or diastolic over 89 mm Hg)
* Have a history of neurological, vascular or psychiatric illness including epilepsy or seizures (excluding depressive illness and anxiety)
* Have a current diagnosis of anxiety or depression
* Are pregnant, trying to get pregnant or breast feeding
* Have a recent history of (within 12 months of screening visit) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as more than 60g (men) / 40g (women) pure alcohol per day (7 / 5.5 units)
* Are (or are seeking to become) pregnant or are lactating
* Have learning difficulties, dyslexia or colour blindness
* Have visual impairment that cannot be corrected with glasses or contact lenses
* Have frequent migraines that require medication (more than or equal to 1 per month)
* Have disorders of the blood
* Have a heart disorder or a history of vascular illness
* Have a respiratory disorder that requires regular medication (Note: participants with asthma who only take their medication occasionally/as required are eligible for this study)
* Have type I or type II diabetes
* Have a history of renal or hepatic disease, or other severe diseases of the gastrointestinal tract (e.g. iron accumulation, iron utilization disorders, hypercalcaemia, hypercalciuria), that are likely to interfere with metabolism/absorption/secretion of the product under investigation
* Have any health condition that would prevent fulfillment of the study requirements
* Are currently or have in the past 4 weeks participated in other clinical or nutrition intervention studies
* Do not have a bank account (required for payment)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function and fatigue during extended performance of the Cognitive Demand Battery (CDB) at 1, 3 and 6 hours post consumption Change in long term declarative memory at 1, 3 and 6 hours post-intervention. | 1-6 hours post intervention

SECONDARY OUTCOMES:
Change in executive function at 1, 3 and 6 hours post intervention. | 1-6 hours post intervention
Change in cerebral blood flow parameters (oxygenated and deoxygenated haemoglobin levels and their sum) in the frontal cortex during task performance commencing at 1, 3 and 6 hours post-intervention. | 1-6 hours post intervention
Change in episodic memory, as measured by immediate word recall, at 1, 3 and 6 hours post intervention. | 1-6 hours post intervention
Change in mood ratings, at 1,3 and 6 hours post intervention. | 1-6 hours post intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, United Kingdom